CLINICAL TRIAL: NCT05635539
Title: A Study of Life Expectancy in Patients With Metabolic Syndrome After Weight Loss: a Comparative Randomized Clinical Trial.
Brief Title: Weight Loss in Patients With COVID-19 and Influenza in Comorbidity With NCDs: a Pilot Prospective Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center, Kazakhstan (Other)
Responsible Party: Principal Investigator, Kuat Oshakbayev, a principal investigator, University Medical Center, Kazakhstan
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AP05135241
Record Dates: First submitted 2022-11-30; First posted 2022-12-02 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Clinical Trial
Keywords: COVID-19; Influenza; Non-Communicable Diseases (NCDs); fast weight loss
MeSH Terms: conditions — COVID-19; Influenza, Human; Noncommunicable Diseases

STUDY DESIGN:
Intervention Model Description: 27 patients with COVID and 35 patients with Influenza
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with COVID (Experimental): 27 patients with COVID in comorbidity with NCDs as T2D, hypertension, and NASH
  Interventions: Dietary Supplement: "Analimentary detoxication" (ANADETO) weight loss based on very-low-calorie-diet
- patients with Influenza (Experimental): 35 patients with Influenza in comorbidity with NCDs as T2D, hypertension, and NASH
  Interventions: Dietary Supplement: "Analimentary detoxication" (ANADETO) weight loss based on very-low-calorie-diet

INTERVENTIONS:
Dietary Supplement: "Analimentary detoxication" (ANADETO) weight loss based on very-low-calorie-diet — calorie restriction to 50-100 kcal/day with fat-free vegetables (tomatoes and cucumbers) with mandatory salt intake to 5-6 gr/day, hot water drinking 1000-1500 ml/day, walking at least 2,000 steps/day after normalized body temperature, and sexual self-restraint. The walking provided to promote of blood circulation and decrease in metabolic intoxication. The weight loss method lasted 14 days. Then the patients followed for 4-week a diet where they ate one meal a day without any food restriction.
  Other Names: very-low-calorie-diet

SUMMARY:
The goal of this study was to evaluate the effects of the fast weight loss on clinic and laboratory inflammation profile, metabolic profile, reactive oxygen species (ROS) and body composition in patients with COVID and Influenza in comorbidity with NCDs.

Primary endpoints: Clinic/infectious/inflammation tests for COVID and Influenza; weight loss during 14 days. Secondary endpoints: fasting blood glucose, HbA1c, blood insulin; systolic/diastolic BP; blood lipids; ALT, AST, chest CT-scan.

DETAILED DESCRIPTION:
Study Design. A 6-week, open, pilot prospective clinical trial with the intention-to-treat principle.

Participants: The study enrolled 72 adult people (38 women) aged from 25 to 80 years with moderate-to-severe cases COVID and Influenza in comorbidity with NCDs as T2D, hypertension, and NASH. All patients with the ARDs had in comorbidity with one or more NCDs. All patients refused for pharmacology therapy due to: either previous unsuccessful drug results; or an antimicrobial resistance profile; or drug allergy; or reluctance to take medication; or iatrogenic fear (iatrophobia); or a rich failed experience in drug treatment; and NASH.

All the patients were admitted into the out-patient department in 3-5 days after illness onset. The study was carried out in the Republic of Kazakhstan from November, 2020, through July, 2022 at University Medical Center (Astana) and ANADETO medical center.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent form;
* patients with fever
* patients refused for pharmacology therapy
* weight loss treatment for 12-14 days and +4 weeks follow-up (total 6 weeks)

Exclusion Criteria:

* patients with acute respiratory failure and assisted ventilation requirement
* respiratory rate ≥ 30 times per minute
* oxygen saturation ≤ 93% by finger oximetry at resting status

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Clinic and infectious tests for COVID and Influenza | Change from Baseline at 6 Weeks
  COVID was diagnosed primarily by direct detection of SARS-CoV-2 RNA by nucleic acid amplification tests with a real-time reverse-transcriptase-polymerase-chain-reaction (RT-PCR) assay. To diagnosis of the flu was used a RT-PCR test called the Flu SC2 Multiplex Assay.
weight loss during 14 days | Change from Baseline at 14 days
  kg
C-reactive protein | Change from Baseline at 6 Weeks
  mg/L

SECONDARY OUTCOMES:
fasting blood glucose | Change from Baseline at 6 Weeks
  mmol/L
glycosylated hemoglobin A1c | Change from Baseline at 6 Weeks
  percent
blood insulin | Change from Baseline at 6 Weeks
  nU/L
systolic/diastolic blood pressures | Change from Baseline at 6 Weeks
  mmHg
blood lipids | Change from Baseline at 6 Weeks
  mmol/L
alanine aminotransferase and aspartate aminotransferase | Change from Baseline at 6 Weeks
  U/L
chest computed tomography scan | Change from Baseline at 14 days
  image

CONTACTS AND LOCATIONS:
Overall Officials: Alaty N Nabiyev, Dr., Study Director — University Medical Center
Locations (1):
- Kuat Pernekulovich Oshakbayev, Astana, Kazakhstan

IPD SHARING:
Plan to Share IPD: No
The investigators will make data available to any investigator/reviewer on their own request, so that the personal privacy of our patients cannot be compromised.

REFERENCES:
- [Derived] Oshakbayev K, Durmanova A, Zhankalova Z, Idrisov A, Bedelbayeva G, Gazaliyeva M, Nabiyev A, Tordai A, Dukenbayeva B. Weight loss treatment for COVID-19 in patients with NCDs: a pilot prospective clinical trial. Sci Rep. 2024 May 14;14(1):10979. doi: 10.1038/s41598-024-61703-1. PMID 38744929